CLINICAL TRIAL: NCT01334853
Title: A Prospective Observational Study to Assess the Role of Selected Biomarkers in Subjects Requiring Daily Medium- to High-dose Inhaled Corticosteroids for Persistent Asthma
Brief Title: A Study to Assess Selected Biomarkers in Subjects Requiring Daily Inhaled Corticosteroids for Persistent Asthma
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MI-CP223
Record Dates: First submitted 2011-03-28; First posted 2011-04-13 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: 50 eosinophilic subjects to be evaluated
  Interventions: Other: No drug will be used
- Cohort 2: 50 non-eosinophilic subjects to be evaluated
  Interventions: Other: No drug will be used

INTERVENTIONS:
Other: No drug will be used — Biomarker
  Groups: Cohort 1
Other: No drug will be used — Biomarker
  Groups: Cohort 2

SUMMARY:
The rationale for conducting this study is to explore potential clinical and peripheral biomarkers in subjects requiring daily medium to high dose inhaled corticosteroids for persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 75 at the time of screening
* Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* History of physician-diagnosed asthma for at least 12 months prior to screening
* Stable Medium- to high-dose ICS divided twice daily as outlined by the NHLBI Asthma Guidelines, 2007

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator or medical monitor, would interfere with interpretation of subject safety or study results
* Concurrent enrollment in another clinical study
* Use of immunosuppressive medication within 3 months prior to screening
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medications with in 30 days prior to screening or during screning period.
* Receipt of immunoglobulin or blood products within 30 days prior to screening or during the screening period
* Receipt of any investigational non-biological drug therapy within 30 days or 5 half-lives prior to screening whichever is longer; or receipt of any marketed or investigational biologic within 6 months or 5 half-lives prior to screening whichever is longer
* Pregnant, lactating, or breastfeeding woman
* Diagnosis of lung disease other than persistent asthma
* History of smoking ≥10 pack years or any smoking within 12 months prior to screening
* History of active, infectious hepatitis A, B, C or human immunodeficiency virus (HIV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with asthma on stable medium- to high-dose inhaled corticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To identify an optimal prediction rule for classifying sputum eosinophilic and non-eosinophilic asthmatics. | 8 Days
  Variables representing lung function tests, patient reported outcomes, and blood biomarkers will be evaluated singly and in various combinations.

SECONDARY OUTCOMES:
To assess which markers are associated with sputum eosinophils. | 8 Days
  Comparing lung function tests between eosinophilic and non-eosinophilic subjects.
To assess which markers are associated with sputum eosinophils | 8 Days
  Comparing blood biomarkers between eosinophilic and non-eosinophilic subjects
To assess which markers are associated with sputum esonophils | 8 Days
  Comparing sputum biomarkers bewteen eosinophilic and non-eosinophilic subjects
To assess which markers are associated with sputum eosinophils. | 8 Days
  Comparing patient reported outcomes between eosinophilic and non-eosinophilic subjects.
To evaluate transcript expression profiles in whole blood and/or sputum using microarray analyses | 8 Days

CONTACTS AND LOCATIONS:
Overall Officials: David Gossage, M.D., Study Director — MedImmune LLC
Locations (18):
- United States (12):
  - Research Site, Denver, Colorado
  - Research Site, Normal, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Madison, Wisconsin
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec